CLINICAL TRIAL: NCT03979131
Title: Phase II Study of Avelumab Plus Chemotherapy in the Peri-operative Treatment for Patients With Resectable Gastric Cancer (GC) or Gastroesophageal Junction Cancer (GEJC)
Acronym: MONEO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO19001
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized, multicentric phase II clinical trial in subjects with operable gastric or GEJ adenocarcinoma. Tissue biopsies before and after treatment will be required. Blood samples will be required at different points of the treatment for biomarker analyses. Tumor imaging assessments will be performed at baseline, after the neoadjuvant treatment, and after finalizing the adjuvancy with avelumab/FLOT, and every 6 months thereafter to determine response to treatment. Clinical decision making will be based on Investigator assessment of the scans using RECIST v1.1. Safety of avelumab/FLOT will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resectable GC and GEJC+avelumab+FLOT preoperative treatment (Experimental): Peri-operatory treatment consisting of four cycles (each cycle is 14 days) of neoadjuvant chemotherapy (docetaxel, oxaliplatin and fluorouracil/leucovorin) plus avelumab previous to surgery. Surgery is recommended to be scheduled 4 to 6 weeks after the last dose. Afterwards (4 to 10 weeks after surgery), four cycles of adjuvant therapy with the same schema, followed by avelumab up to one year.
  Interventions: Combination Product: Avelumab addition to perioperative chemotherapy in GC and GEJC

INTERVENTIONS:
Combination Product: Avelumab addition to perioperative chemotherapy in GC and GEJC — Avelumab addition to perioperative chemotherapy in GC and GEJC. Peri-operatory treatment consisting of four cycles (each cycle is 14 days) of neoadjuvant chemotherapy (docetaxel, oxaliplatin and fluorouracil/leucovorin) plus avelumab previous to surgery. Surgery is recommended to be scheduled 4 to 6 weeks after the last dose. Afterwards (4 to 10 weeks after surgery), four cycles of adjuvant therapy with the same schema, followed by avelumab up to one year. There will be be a follow-up of 5 years.

SUMMARY:
Phase II Study of Avelumab plus chemotherapy in the peri-operative treatment for patients with resectable Gastric cancer (GC) or Gastroesphageal Junction cancer (GEJC)

The addition of Avelumab to the perioperative chemotherapy in GC and GEJC patients may increase pathological responses by a synergic effect activating the immune response. Conclusively, the survival of these patients would improve.

The primary objective is to investigate whether the addition of avelumab to FLOT chemotherapy (docetaxel, oxaliplatin and fluorouracil/leucovorin) improves efficacy in terms of pathological complete response (pCR) rate, in GC and GEJC patients compared to the historical data of chemotherapy alone in the neoadjuvant setting.

DETAILED DESCRIPTION:
Phase II Study of Avelumab plus chemotherapy in the peri-operative treatment for patients with resectable Gastric cancer (GC) or Gastroesphageal Junction cancer (GEJC)

The addition of Avelumab to the perioperative chemotherapy in GC and GEJC patients may increase pathological responses by a synergic effect activating the immune response. Conclusively, the survival of these patients would improve.

The primary objective is to investigate whether the addition of avelumab to FLOT chemotherapy (docetaxel, oxaliplatin and fluorouracil/leucovorin) improves efficacy in terms of pathological complete response (pCR) rate, in GC and GEJC patients compared to the historical data of chemotherapy alone in the neoadjuvant setting.

Secondary objectives are as follows:

* To evaluate the addition of avelumab to the perioperative chemotherapy in regard to the following:

  * Overall survival (OS)
  * Disease-free survival (DFS)
  * Progression-free survival (PFS)
  * Surgical resection rate (R0)
  * Overall Response Rate (ORR) to neoadjuvancy
* To determine the safety and tolerability of avelumab with FLOT chemotherapy.
* To perform a comprehensive analysis of biomarkers, as exploratory endpoints.

Study design: This is an open-label, non-randomized, multicentric phase II clinical trial in subjects with operable gastric or GEJ adenocarcinoma. Tissue biopsies before and after treatment will be required. Blood samples will be required at different points of the treatment for biomarker analyses. Tumor imaging assessments will be performed at baseline, after the neoadjuvant treatment, and after finalizing the adjuvancy with avelumab/FLOT, and every 6 months thereafter to determine response to treatment. Clinical decision making will be based on Investigator assessment of the scans using RECIST v1.1. Safety of avelumab/FLOT will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported.

Study population: Patients with resectable gastric and GEJ cancer suitable for preoperative chemotherapy.

Statistical Considerations: Summary tables (descriptive statistics and frequency tables) will be provided for all demographic, baseline and safety variables, as appropriate. Continuous variables will be summarized with descriptive statistics (mean, standard deviation, range, and median). Ninety-five (95) percent confidence intervals (95% CI) may also be presented, as appropriate. Frequency counts and percentage of subjects within each category will be provided for categorical data. The primary efficacy analysis (pCR) will be performed using the binomial test procedure. Additionally, for the pCR rate one-sided 90% CI will be also presented to be consistent with sample size calculation. Secondary endpoints will be summarized with descriptive statistics. Survival analysis will be performed to analyse OS, PFS and DFS. Kaplan- Meier curves will be presented and possible comparisons will be tested using the log-rank test or the Cox proportional hazard model for multivariate analysis, hazard ratios (HR) and their 95% confidence interval (CI95%) will be provided. Any survival analyses will be considered as exploratory.

The study population are patients with resectable gastric and GEJ cancer suitable for preoperative chemotherapy. The study duration will be approximately 24 months of recruitment; 5 years of additional followup.

Regarding to the study product, peri-operatory treatment consisting of four cycles (each cycle is 14 days) of neoadjuvant chemotherapy (docetaxel, oxaliplatin and fluorouracil/leucovorin) plus avelumab previous to surgery. Surgery is recommended to be scheduled 4 to 6 weeks after the last dose. Afterwards (4 to 10 weeks after surgery), four cycles of adjuvant therapy with the same schema, followed by avelumab up to one year.

Finally, this study will be conducted in 10 centres in Spain.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven, gastric or GEJ adenocarcinoma (Siewert I-III).
2. Availability of a paraffin block from the diagnostic endoscopic biopsy (and a fresh biopsy if possible), and a second tumor block (fresh + paraffin) from the surgical specimen.
3. Have evaluable disease as defined by RECIST 1.1 and determined by investigator assessment, with the absence of distant metastases on CT scan of thorax, abdomen and pelvis.
4. Patient medically fit and amenable to gastrectomy/esophagectomy with curative intent as confirmed by a multidisciplinary team discussion.
5. UICC tumor stage Ib (T1N1 only, T2N0 not eligible) to IIIC, as defined by CT, according to the 7th AJCC Edition.
6. Age ≥ 18 years.
7. WHO performance status 0-1.
8. Adequate organ function (assessed within 7 days prior treatment initiation):

   1. White blood cell count (WBC) > 3 x 109 /L
   2. Absolute neutrophil count (ANC) > 1.5 x 109 /L
   3. Platelets ≥ 100 x 109 /L
   4. Estimated glomerular filtration rate should be > 50 ml/min
   5. Total bilirubin within normal limits (if the patient has documented Gilbert's disease ≤ 1.5 x ULN or direct bilirubin ≤ ULN).
   6. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN.
9. In case of anticoagulation, investigator and patient should agree to replace any oral anticoagulation by subcutaneous administration of low-molecular weight heparin in equivalent doses before treatment start;
10. For women who are not postmenopausal (> 12 months of non-therapy induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last treatment dose.
11. For men: agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last dose of study treatment. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods for contraception.
12. For all female patients who are not confirmed postmenopausal (> 12 months of non-therapy induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus) a negative serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) result should be available before treatment and within 7 days from treatment start should be performed. Female patients should not be breast feeding.
13. Written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

1. Other histology different from adenocarcinoma.
2. Has had previous therapy for gastric or GEJ cancer.
3. Known hypersensitivity to the components of anti-PD-L1, docetaxel, oxaliplatin, fluorouracil/leucovorin.
4. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
5. Previous malignancy within the last 5 years, except for adequately treated cervical carcinoma in situ, localized non-melanoma skin cancer, or other curatively treated cancer without impact on the patient's overall prognosis according to the judgment of the investigator.
6. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those condition should be discussed with the patient before registration in the trial.
7. History of clinically significant comorbidities.
8. Patients medically unfit for FLOT chemotherapy, according to the local guidance.
9. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxin, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication). History or evidence of interstitial lung disease or active, non-infectious pneumonitis.
11. Active infection requiring systemic therapy.
12. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or Active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected). Test for HBV and HCV are required for the screening.
13. Received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu-vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.
14. Prior organ transplantation including allogenic stem-cell transplantation.
15. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI-CTCAE v4.0 Grade ≥ 3).
16. Persisting toxicity related to prior therapy (NCI-CTCAE v4.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
17. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
18. Pregnant women and lactating females are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 7 years
  Pathological complete response (pCR) rate, where pCR is defined as the absence of residual tumor based on evaluation of the resected esophagogastric specimen according to Becker remission criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 7 years
  Overall survival (OS) [time frame: from the initial date of neoadjuvant chemotherapy to the date of death due to any cause. Patients without documentation of death at the time of analysis will be censored at the last follow-up date]. Estimated using Kaplan-Meier method.
Disease-free survival (DFS) | 7 years
  Disease-free survival (DFS) [time frame: from the surgery to the first observation of disease relapse or death due to any cause. Patients without an event prior to the time of analysis will be censored at the last relapse free assessment]. Relapse is defined according to RECIST v1.1. Estimated using Kaplan Meier method.
Progression-free survival (PFS) | 7 years
  Progression-free survival (PFS) [time frame: from the initial date of neoadjuvant chemotherapy to the date of first documentation of disease progression or death due to any cause, whichever occurs first. Patients without an event prior to the time of analysis will be censored at the last assessment that is stable disease (SD) or better]. Progression is defined according to RECIST v1.1. Estimated using Kaplan-Meier method.
Surgical complete resection rate (R0) | 2 years
  Surgical complete resection rate (R0). This is a complete macroscopic resection of the gross tumor with negative surgical margins

CONTACTS AND LOCATIONS:
Overall Officials: María Alsina Maqueda, PhD, Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (1):
- Vall d'Hebron Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069